CLINICAL TRIAL: NCT03932526
Title: Combined Use of Apatinib Mesylate and Vinorelbine Versus Single Use of Vinorelbine in Recurrent or Metastatic Triple-negative Breast Cancer: a Double-blinded Randomized Controlled Clinical Trial
Brief Title: Combined Use of Apatinib Mesylate and Vinorelbine Versus Single Use of Vinorelbine in Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Sun Tao, Department director, Liaoning Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STao-003
Record Dates: First submitted 2019-04-15; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Vinorelbine; apatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinorelbine + placebo group (Active Comparator): 92 enrolled patients will be assigned to receive oral vinorelbine plus placebo until disease progression or other criteria for administration termination.
  Interventions: Drug: Vinorelbine + placebo
- Vinorelbine + Apatinib group (Experimental): 92 enrolled patients will be assigned to receive oral patatinib mesylate in combination with vinorelbine until disease progression or other criteria for administration termination.
  Interventions: Drug: Vinorelbine + Apatinib

INTERVENTIONS:
Drug: Vinorelbine + placebo — Combined administration of vinorelbine and placebo. Based on oral administration of vinorelbine, the patients will be given oral placebo (starch as an ingredient). The placebo appearance, including shape, size, color and weight, taste, labeling and packing are the same with those of apatinib mesylate tablets.
  Other Names: AiTan+ placebo
  Arms: Vinorelbine + placebo group
Drug: Vinorelbine + Apatinib — Combined administration of vinorelbine and apatinib. Vinorelbine tartrate soft capsule (also named Navelbine; registration No. H20140657; Pierre Fabre Medicament, Boulogne, France) 40 mg once orally, taken in the morning (at least 1 hour before or at least 1 hour after meals), three times a week (Mondays, Wednesdays, and Fridays), for a continuous 21-day cycle. Apatinib mesylate tablets (also named Aitan, State Medical Permission No. H20140103; Jiangsu Hengrui Pharmaceutical Co., Ltd., China), 500 mg orally, taken once a day for a continuous 21-day cycle.
  Other Names: Navelbine+AiTan
  Arms: Vinorelbine + Apatinib group

SUMMARY:
To compare the therapeutic effect of vinorelbine used alone or combined with apatinib mesylate for recurrent or metastatic TNBC patients who have at least received one chemotherapy regimen, including anthracyclines and taxanes, providing clinical evidence for multi-line treatment options for advanced TNBC.

DETAILED DESCRIPTION:
The emergence of new molecular targeted drugs provides new prospects for the treatment of advanced breast cancer; and its future therapeutic trend includes chemotherapy combined with molecular targeted therapy. Apatinib mesylate (Aitan), a novel small molecule anti-angiogenic agent, highly selectively inhibits the activity of vascular endothelial growth factor receptor-2 tyrosine kinase. Aitan also blocks the signaling of vascular endothelial growth factor binding to its receptor, thereby strongly inhibiting tumor angiogenesis and exerting anti-tumor effect.However, a randomized controlled clinical trial of apatinib combined with vinorelbine for TNBC has not been reported. The objective of this study is to compare the therapeutic effect of vinorelbine alone or combined with apatinib mesylate for recurrent or metastatic triple-negative breast cancer (TNBC) patients who have received at least two regimens containing anthracyclines and taxanes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with recurrent or metastatic TNBC, as confirmed by histological or cytological examination
* Age 18-70 years old
* According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, there is at least one measurable lesion.
* The Eastern Cooperative Oncology Group (ECOG) scores 0-2
* Expected survival ≥ 12 weeks
* Negative for ER/PR
* All patients will be tested for bone marrow capacity, liver and renal functions within 7 days prior to enrollment
* Previous use of anthracyclines and/or taxanes
* The medication history of vinorelbine
* Female patients of childbearing age must take adequate contraception; otherwise the patients must be proven to be infertile
* No history of serious heart, lung, liver, and kidney diseases
* Provision of written informed consent

Exclusion Criteria:

* Patients who receive chemotherapy, radiation therapy, targeted drugs, or hormone therapy within 3 weeks of administration
* Patients using corticosteroids for untreated brain or subdural metastatic lesions, need to have stopped it, at least for 4 weeks or until there are no signs of brain metastasis and/or symptoms must have stabilized for at least 4 weeks, if local treatment has been completed. Enhanced computed tomography (CT) or magnetic resonance imaging (MRI) images during screening are compared with those performed at least 4 weeks earlier to determine radiological stability.
* Patients with severe vascular diseases, including unstable angina, myocardial infarction, or severe arrhythmia in the past 6 months
* History of HIV infection or active chronic hepatitis B or C
* Patients with other serious infectious diseases
* Patients positive for ER/PR/HER-2 positive
* Patients with allogeneic organ transplants requiring immunosuppressive therapy
* History of other malignant tumors within 5 years, except for cured cervical carcinoma in situ or basal cell carcinoma of the skin
* Other destabilizing factors that may interfere with patients or have an impact on the trial results
* Allergic to target drugs or allergic to related drugs applied in the trial
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2019-06-24 (Estimated); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-06-26 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival(PFS) | Day 1 of treatment until disease progression or death from any cause, assessed up to 24 months
  PFS refers to the length of time from random enrollment to any recorded tumor progression or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months
  OS indicates the length of time from enrollment to death from any cause.When no information on death is collected in the clinical database, the last date when the patient is still known to have survived is used as the cut-off point.
Disease control rate (DCR) | Up to 24 months
  DCR indicates the percentage of patients with CR, partial remission, and disease stabilization; and maintenance over 4 weeks, accounts for all the subjects with evaluable efficacy.
Overall remission rate (ORR) | Up to 24 months
  ORR is the proportion of patients who achieve a complete or partial response ((CR+PR)/total number of cases x 100%), as assessed by the RECIST v1.1.
Adverse events at levels 3 and 4 | every 6 weeks (two cycles) and 4 weeks after treatment discontinuation
  Patients with adverse events at levels 3 and 4 will be assessed according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Sun, Principal Investigator — Liaoning Cancer Hospital & Institute

REFERENCES:
- [Derived] Wu S, Zhang L, Li H, Xu J, Jiang C, Sun T. Combined use of apatinib mesylate and vinorelbine versus vinorelbine alone in recurrent or metastatic triple-negative breast cancer: study protocol for a randomized controlled clinical trial. Trials. 2020 May 24;21(1):420. doi: 10.1186/s13063-020-04342-x. PMID 32448335